CLINICAL TRIAL: NCT06537466
Title: A Randomised Controlled Tria of Low-calorie Ketogenic Diet Versus Mediterranean Diet in Patients With Compensated Advanced Chronic Liver Disease (cACLD) Secondary to Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Brief Title: Ketogenic Diet in MASLD-related cACLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Salvatore Petta, Associate Professor of Gastroenterology, MD, PhD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KETOMASH
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Steatohepatitis, Nonalcoholic; Steatosis of Liver; Cirrhosis, Liver
Keywords: Steatohepatitis; Steatosis; Ketogenic diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Active Comparator): This equilibrated diet has a caloric value 10% below the total metabolic expenditure of each individual. The total metabolic expenditure is calculated from the basal metabolic expenditure (based on the formula FAO/WHO/UN) multiplied by the coefficient of activity, which is calculated according to the physical activity of each participant. The calories provide to this group range between 1,400 and 1,800 kcal/day. The ration of macronutrients provided is 45-55 % arbohydrates,15-25 % proteins, and 25-35 % fat, in addition to a recommended intake of 20-40 g/day of fiber in the form of vegetables and fruits.
  Interventions: Dietary Supplement: Mediterranean diet
- Very Low Ketogenic Diet (Experimental): The VLCKD ketogenic protocol entails: a caloric intake < 800 calories, a protein intake calculated based on individual needs: 1.2 + 0.2 g/kg/ideal body weight, low carbohydrate content (approximately 45-55 g of carbohydrates per day), and low lipids (10-15g/day). Vitamins and minerals, Unlimited vegetables.
  Interventions: Dietary Supplement: Very Low Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — This equilibrated diet has a caloric value 10% below the total metabolic expenditure of each individual. The total metabolic expenditure is calculated from the basal metabolic expenditure (based on the formula FAO/WHO/UN) multiplied by the coefficient of activity, which is calculated according to the physical activity of each participant. The calories provide to this group range between 1,400 and 1,800 kcal/day. The ration of macronutrients provided is 45-55 % arbohydrates,15-25 % proteins, and 25-35 % fat, in addition to a recommended intake of 20-40 g/day of fiber in the form of vegetables and fruits.
  Arms: Mediterranean Diet
Dietary Supplement: Very Low Ketogenic Diet — The VLCKD ketogenic protocol entails: a caloric intake < 800 calories, a protein intake calculated based on individual needs: 1.2 + 0.2 g/kg/ideal body weight, low carbohydrate content (approximately 45-55 g of carbohydrates per day), and low lipids (10-15g/day). Vitamins and minerals, Unlimited vegetables.
  Arms: Very Low Ketogenic Diet

SUMMARY:
The investigators hypothesize that very low ketogenic diet could represent a new therapeutic option in the management of patients with MASLD and cACLD. Therefore, the investigator propose a randomized controlled study that evaluates the impact of two dietary protocols -Mediterranean diet, and very low ketogenic diet- the MD and the VLCKD, in individuals with cACLD secondary to MASLD.

DETAILED DESCRIPTION:
The rationale of the study stems from evidence that patients with "compensated advanced chronic liver disease" (cACLD) secondary to MASLD have higher risk of liver-related morbidity (liver decompensation, hepatocellular carcinoma) and mortality. However, todate the only approved drug by FDA in patients with MASH and F2-F3 fibrosis is Resmetirom, but it is still not available in clinical practice outside US. As a consequence, currently and in the future the first-line treatment of MASLD involved weight loss and lifestyle modification, such as physical exercise and dietary regimens based on calorie restriction. In this context the Mediterranean diet is considered the standard, but over the last decade, the Very low-carbohydrate ketogenic diets (VLCKD) has gained immense popularity for its short-term positive effects on weight loss, even if data on MASLD cACLD are lacking.

Therefore, considering recent evidence, the investigator hypothesize that VLCKD could represent a new therapeutic option in the management of patients with MASLD and cACLD. Specifically, the investigator propose a randomized controlled study that evaluates the 48 week impact of two dietary protocols, the MD and the VLCKD, in individuals with cACLD secondary to MASLD, with specific focus on weight loss >=10% and on liver-related (changes in liver stiffness by TE, MRE and MRI-PDFF, AST, ALT) and metabolic parameters (see section on outcomes) Here the investigators report the detailed proposed nutritional protocols

* MEDITERRANEAN DIET This equilibrated diet has a caloric value 10% below the total metabolic expenditure of each individual. The total metabolic expenditure is calculated from the basal metabolic expenditure (based on the formula FAO/WHO/UN) multiplied by the coefficient of activity, which is calculated according to the physical activity of each participant. The calories provide to this group range between 1,400 and 1,800 kcal/day. The ration of macronutrients provided is 45-55 % arbohydrates,15-25 % proteins, and 25-35 % fat, in addition to a recommended intake of 20-40 g/day of fiber in the form of vegetables and fruits.
* VERY LOW-CARBOHYDRATE KETOGENIC DIETS The VLCKD ketogenic protocol entails: a caloric intake < 800 calories, a protein intake calculated based on individual needs: 1.2 + 0.2 g/kg/ideal body weight, low carbohydrate content (approximately 45-55 g of carbohydrates per day), and low lipids (10-15g/day). Vitamins and minerals, Unlimited vegetables.

The Kalibra protocol consists of 3 stages:

WEIGHT LOSS: Ketogenic metabolism is activated by reduced carbohydrate intake. As an accessory phenomenon to lipolysis and the catabolism of fat reserves in adipose tissue, there is a physiological production of ketone bodies (acetoacetate, beta-hydroxybutyrate, acetone), which represent a water-soluble and readily available energy source for many tissues in the body (brain, heart, and muscles). Continuous ketogenesis, in addition to providing adequate energy intake, is important to ensure the absence of hunger and a feeling of overall well-being throughout the weight loss period.

TRANSITION: gradual reintroduction of traditional foods. In this phase, the patient is reeducated to adopt a healthy and correct lifestyle in order to optimize and stabilize the results obtained in the attack phase.

MAINTENANCE: once the patient has achieved their overall goals, they embark on a long-term nutritional path following the LARN (Reference Intake Levels of Nutrients and Energy for the Italian population).

In the first phase, known as the classic ketogenic phase (21 days), the protocol involves replacing all meals with Kalibra products, accompanied by low-carbohydrate vegetables. It is essential to include supplementation with trace elements, minerals, and vitamins. The number of meals is determined based on the patient's height in centimeters (tab1).

During the period when following the Kalibra method, it is recommended to engage in physical activity for muscle toning of arms, legs, abdominals, and glutes for 20-30 minutes at least 3 times a week. A workout plan will be provided.

Table 1 height in centimeters <160 160-170 170-180 >180 Man 3-4 meals 4 meals 4-5 meals 5 meals Woman 5 meals 5 meals 6 meals 6-7 meals Tab1 Number of meal replacements based on height. The second ketogenic phase, called the Mitigated Diet (21 days), involves reducing one Kalibra meal and the possibility of adding a portion of meat, fish, or eggs during one of the main meals, accompanied by low-carbohydrate vegetables. This allows for the maintenance of ketogenesis with consequent weight loss while also allowing the patient a reasonable level of social interaction.

The Transition Phase represents an extremely important phase as it allows for the stabilization of the achieved weight through a gradual and measured increase in daily caloric intake.

Each stage, each lasting 21 days, involves a caloric increase of approximately 150 kcal correlated with:

* Gradual numerical reduction of Kalibra protein foods
* Increase in carbohydrate intake using low glycemic index foods
* Introduction of foods from the Mediterranean diet
* Progressive reduction of micronutritional supplementation The gradual caloric increase, carried out in each of the 4 stages of the transition phase, allows for the stabilization of the weight achieved with the Kalibra Method and its maintenance in the long term.

Once the 4 stages of the transition are completed, the patient will have finished their dietary journey and can then maintain the achieved results by daily application of a new lifestyle based on healthy and balanced nutrition, taking into account fundamental aspects of the Mediterranean diet.

* Consume at least five servings of fruits and vegetables as they are rich in fiber, vitamins, minerals, and antioxidant substances.
* Maintain proper hydration levels by consuming at least 1.5-2 liters of water per day.
* Start the day with a balanced breakfast to keep key hunger-regulating mechanisms in check, resulting in reduced hunger throughout the day.
* Distribute daily caloric intake into at least four meals, preferably adhering to the following percentages: breakfast 27%, lunch 36%, snack 13%, and dinner 24%.
* Consume foods with a low glycemic index and load.

Here the investigators report the detailed clinical and laboratory assessment:

Nutritional status will be assessed using the Royal Free Hospital-Nutritional Prioritizing Tool (RFH-NPT), recommended by the European Society for Clinical Nutrition and Metabolism (ESPEN) guidelines for stratifying malnutrition risk in patients with liver diseases. Evaluation will include: Weight (Kg), height (cm), waist and hip circumference (cm), arm circumference (cm), triceps skinfold (using a caliper), thigh and suprapatellar root measurements. Body mass index (BMI) will be calculated based on weight in kilograms and height in meters.

Body composition will be assessed using bioimpedance analysis and muscle strength will be evaluated using a dynamometer. A walking test will be conducted, and the Liver Frailty Index will be calculated.

Weight and circumferences will be assessed at each visit. A comprehensive evaluation will be performed at the end of each phase.

A 12-hour overnight fasting blood sample will be drawn at screening and during follow-up visits determine serum levels of Hb, WBC, ALT, AST, ɣ-glutamyltransferase (ɣ-GT) , alkaline phosphatase, total and direct bilirubin, INR, albumin, total cholesterol, HDL and LDL-cholesterol, triglycerides, plasma glucose concentration, platelet count , NA/K and creatinine.

Here the investigators report the detailed liver instrumental assessment:

At baseline, all patients will undergo an ultrasound (US) examination to evaluate liver structure and the presence of signs of portal hypertension. Transient elastography will be performed using a FibroScan apparatus (Echosens, Paris , France) to measure liver stiffness and controlled attenuation parameter. The median value of 10 successful acquisitions, expressed in kilopascal (kPa), will be kept as representative of LSM. The investigator will consider 10 successful acquisitions with a success rate of at least 60% and with an interquartile range lower than 20% as representative measurements. During the same session, MRE and MRI-PDFF will be used as diagnostic tools for noninvasive quantitative assessment of steatosis and liver fibrosis; muscle mass will be also evaluated at L3 level. Transient elastography will be repeated every three months, US will be repeated every six months, and the MRE and MRI-PDFF will be performed at the end of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years
2. Pattients with cACLD secondary MASLD. Specifically cACLD is defined as liver stiffness ≥10 KPa by Transient Elastography and/or fibrosis F3 or F4 at liver biopsy by Kleiner scoring system; MASLD is defined by the presence of steatosis and at least one of five cardiometabolic risk factor.
3. Informed consent form obtained before any trial-related ac.vity.

Exclusion Criteria:

1. Concomitance of any other chronic liver disease: Wilson's disease (normal serum ceruloplasmin); alpha-1-an.trypsin deficiency (normal serum alpha-1-an.trypsin); viral hepatitis (anti-HCV and HBsAg negativity); primary biliary cirrhosis (ANA<1:160 and AMA negativity); autoimmune hepatitis (ANA, SMA and LKM <1:160), . .
2. MetALD: patients with metabolic dysfunc.on-associated steato.c liver disease, who consume amounts of alcohol per week (140-350 g/wk and 210-420 g/wk for females and males, respectively.
3. History of or planned gastrointestinal bypass or any additional bariatric surgery/intervention.
4. Recent significant weight loss ( > 5 % within previous 6 months)
5. Presence of large esophageal varices (F2 or F3)
6. Decompensated liver cirrhosis and/or presence of hepatocarcinoma and/or portal thrombosis.
7. Be pregnant or breasxeeding.
8. Type 1 diabetes, cardiac arrhythmias, recent stroke or myocardial infarction, heart failure, elective surgery or invasive procedures, chronic kidney disease (eGFR<30 ml/min).
9. Therapy with SGLT-2 inhibitors and/or GLP-1 agonist started within 6 months of screening visit.
10. Recent (within 6 months of screening visit) or concomitant use of agents known to cause hepatic steatosis (corticosteroids, amiodarone, methotrexate, tamoxifen, tetracycline, high dose estrogens, valproic acid)
11. Any additional condition that might interfere with optimal participation in the study, according to investigators opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
weight loss≥10% compared to the initial weight in individuals with cACLD secondary to MASLD | 48 weeks
  Weight in Kg

SECONDARY OUTCOMES:
▪ changes in liver stiffness by Magnetic Resonance Elastography (MRE) | 48 weeks
  MRE in KPa
▪ changes in liver fat by Magnetic Resonance Imaging-proton density fat fraction (MRI-PDFF) | 48 weeks
  MRI-PDFF in %
▪ changes in liver stiffness by transient elastography | 48 weeks
  Liver Stiffness in KPa
▪ changes in liver fat by controlled attenuation parameter (CAP) | 48 weeks
  CAP in dB/m
▪ changes in Spleen stiffness by Magnetic Resonance Elastography (MRE) | 48 weeks
  Spleen Stiffness in KPa
▪ changes in Spleen stiffness by Transient Elastography | 48 weeks
  Spleen stiffness in KPa
▪ changes in AST serum levels | 48 weeks
  AST in IU
▪ changes in ALT serum levels | 48 weeks
  ALT in IU
▪ changes in GGT serum levels | 48 weeks
  GGT in IU
▪ changes in alcaline phosphatase serum levels | 48 weeks
  alcaline phosphatase in IU
▪ changes in albumin serum levels | 48 weeks
  albumin in g/L
▪ changes in INR serum levels | 48 weeks
  INR in IU
▪ changes in bilirubin serum levels | 48 weeks
  bilirubin in mg/dl
▪ changes in total, HDL and LDL cholesterol serum levels | 48 weeks
  total, HDL and LDL cholesterol in mg/dl
▪ changes in glucose serum levels | 48 weeks
  gluceos in mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Gastroenterology, PROMISE, University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No